CLINICAL TRIAL: NCT02911142
Title: Phase I/II Study of Lenalidomide Combined With Modified DA-EPOCH and Rituximab (EPOCH-R2) in Primary Effusion Lymphoma or KSHV-Associated Large Cell Lymphoma
Brief Title: Lenalidomide Combined With Modified DA-EPOCH and Rituximab (EPOCH-R2) in Primary Effusion Lymphoma or KSHV-associated Large Cell Lymphoma
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ramya Ramaswami, Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 160171; 16-C-0171
Record Dates: First submitted 2016-09-21; First posted 2016-09-22 (Estimated); Results first posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Primary Effusion Lymphoma; B-Cell Neoplasm
Keywords: Treatment Naive; Immune Modulatory; Chemotherapy; AIDS-Related Lymphoma; PEL
MeSH Terms: conditions — Lymphoma, Primary Effusion; Lymphoma, B-Cell; Lymphoma, AIDS-Related | interventions — Lenalidomide; Rituximab; Prednisone; Etoposide; etoposide phosphate; Doxorubicin; liposomal doxorubicin; Vincristine; Cyclophosphamide; Electrocardiography; Echocardiography; Ultrasonography; Bronchoscopy; Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lenalidomide, Rituximab, Prednisone, Etoposide, Doxorubicin, Vincristine and Cyclophosphamide (Experimental): Lenalidomide, Rituximab, Prednisone, Etoposide, Doxorubicin, Vincristine and Cyclophosphamide
  Interventions: Drug: Lenalidomide; Drug: Rituximab; Drug: Prednisone; Drug: Etoposide; Drug: Doxorubicin; Drug: Vincristine; Drug: Cyclophosphamide; Diagnostic Test: CT of neck, chest, abdomen and pelvis; Diagnostic Test: 18FDG-PET scan; Diagnostic Test: MRI Brain; Procedure: Bone marrow biopsy; Diagnostic Test: EKG; Diagnostic Test: Echocardiogram; Diagnostic Test: Ultrasound; Diagnostic Test: Bronchoscopy; Diagnostic Test: Endoscopy; Diagnostic Test: CXR: PA/lat/decub

INTERVENTIONS:
Drug: Lenalidomide — Lenalidomide taken orally, daily at assigned dose level on days 1 to 10, up to 25mg.
  Other Names: Revlimid
Drug: Rituximab — During cycle 1, rituximab will be administered on day 4 prior to the start of etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin (EPOCH). During cycles 2 to 6, rituximab will be administered on day 1 of each cycle.
  Other Names: Rituxan; Riabni; Ruxience; Truxima
Drug: Prednisone — During cycle 1, Prednisone 60 mg/m^2 /day by mouth (PO) days 6 to 10. During cycles 2-6, Prednisone 60 mg/m^2 /day PO days 1-5.
  Other Names: Rayos; Deltasone; Prednisone Intensol
Drug: Etoposide — During cycle 1, Etoposide 50 mg/m^2 /day continuous intravenous infusion days 6 to 9. During cycles 2-6, Etoposide 50 mg/m^2/day continuous intravenous infusion days 1 to 4.
  Other Names: Toposar; Etopophos
Drug: Doxorubicin — During cycle 1, Doxorubicin 10 mg /m^2/day continuous intravenous infusion days 6 to 9. During cycles 2-6, Doxorubicin continuous intravenous infusion days 1 to 4.
  Other Names: Lipodox; Lipodox 50; Doxil
Drug: Vincristine — During cycle 1, Vincristine 0.4 mg/m^2 /day continuous intravenous infusion days 6 to 9. During cycles 2-6, Vincristine continuous intravenous infusion days 1 to 4.
  Other Names: Oncovin; Marqibo; Vincasar PFS
Drug: Cyclophosphamide — During cycle 1, Cyclophosphamide 750 mg/m^2 day 10. During cycles 2-6, Cyclophosphamide 750 mg/m^2 day 5.
  Other Names: Cytoxan; Neosar; Endoxan
Diagnostic Test: CT of neck, chest, abdomen and pelvis — Screening
  Other Names: Computed tomography of neck, chest, abdomen and pelvis
Diagnostic Test: 18FDG-PET scan — Baseline
  Other Names: 18 F-fluorodeoxyglucose-positron emission tomography scan
Diagnostic Test: MRI Brain — Screening
  Other Names: Magnetic resonance imaging brain
Procedure: Bone marrow biopsy — Baseline
  Other Names: BM biopsy
Diagnostic Test: EKG — Screening
  Other Names: electrocardiogram
Diagnostic Test: Echocardiogram — Screening
  Other Names: ECHO
Diagnostic Test: Ultrasound — Day 6
  Other Names: U/S
Diagnostic Test: Bronchoscopy — Baseline
Diagnostic Test: Endoscopy — Baseline
Diagnostic Test: CXR: PA/lat/decub — Screening
  Other Names: Chest x-ray posteroanterior, lateral, decubitus

SUMMARY:
Background:

Primary effusion lymphoma (PEL) is a rare disease with no standard treatment. Researchers want to see if a drug called lenalidomide along with common chemotherapy drugs may be effective in treating PEL.

Objective:

To test a new treatment for PEL.

Eligibility:

People ages 18 and older with PEL.

Design:

Participants will be screened with blood tests, imaging studies, a physical exam, and other tests.

Participants will have tests to evaluate their disease. These may include:

Blood tests

Scans

Lumbar puncture. Fluid around the spinal cord will be removed with a needle.

Bone marrow removed with a needle and studied

Samples of skin or lymph nodes removed

Fluid removed from around organs

Lung and eye tests

Tubes with cameras taking pictures of airways or digestive tract

Participants will take lenalidomide pills for 10 days. They will keep a pill diary.

Participants will have a catheter (small tube) placed in the large vein in the arm or chest.

Participants will get DA-EPOCH-R as intravenous infusions by catheter over several days. This will be repeated in 21-day cycles. Most participants will have 6 cycles.

Participants will get the drug filgrastim by injection under the skin. They will get the drug methotrexate injected into the spinal fluid.

During the study, participants will have the following tests done at least once:

Medical history

Physical exam

Blood, urine, and stool tests

Lesions photographed and measured

Lumbar puncture

Participants will have follow-up visits for 5 years. They will repeat the screening tests plus have urine and stool tested.

Participants may be contacted later by phone to see how they are doing.

DETAILED DESCRIPTION:
Background

* Kaposi sarcoma herpesvirus (KSHV)-associated primary effusion lymphoma (PEL) is an aggressive B cell neoplasm with clinicopathologic and molecular profiles distinct from other AIDS-related lymphomas.
* There are no prospective studies on these rare lymphomas. Clinical experience is limited; however, reported prognosis is poor, with median survival estimated at less than 6 months using conventional cyclophosphamide, doxorubicin, vincristine, prednisone (CHOP)-like chemotherapy.
* Novel treatment is urgently needed for KSHV-associated lymphomas, and the therapeutic approach must take into account concurrent KSHV-associated malignancies which are commonly seen in this patient population
* Lenalidomide, an immune-modulatory derivative of thalidomide (IMiD drug) has in vitro direct antitumor effect in KSHV-lymphomas as well as immune modulatory and anti-angiogenic effects that may be beneficial in treating PEL.
* Rituximab, an anti-cluster of differentiation 20 (CD20) monoclonal antibody, has recently been shown to be an active agent in the management of KSHV-MCD. Although PEL is a CD20-negative tumor, advances in the understanding the biology of KSHV-infection of B-cells, the pathobiology of IL-6 syndromes in KSHV-Multicentric Castleman disease (MCD) and KSHV-non-Hodgkin lymphoma (NHL), and clinical experience using rituximab in the treatment of KSHV-MCD, support use of rituximab in the treatment of PEL, especially in patients with concurrent KSHV-MCD.
* Modified dose-adjusted etoposide, prednisone, vincristine, cyclophosphamide, and doxorubicin (DA)-EPOCH is an anthracycline-based regimen that allows for personalization of dose-intensity showing that inclusion of etoposide and infusional administration decreases tumor cell resistance.
* The use of DA-EPOCH in combination with rituximab for the treatment of human immunodeficiency virus (HIV) associated diffuse large B-cell lymphoma or Burkitt lymphoma has been shown to be safe and effective.
* Given the central role of controlling HIV viremia with combination antiretroviral therapy (cART) in the management of KSHV-associated malignancies, as well as the likely contribution of uncontrolled HIV viremia to PEL pathogenesis, cART will be employed as an important part of the treatment regimen.

Objectives

Phase I

- Evaluate safety and tolerability of lenalidomide in combination with DA-EPOCH-R and determine the maximum tolerated dose and/or recommended phase II dose of this regimen.

Phase II

- Evaluate overall survival in treatment-naive participants with KSHV-positive aggressive B cell lymphomas treated with lenalidomide in combination with DA-EPOCH and rituximab (DA-EPOCH-R^2).

Eligibility

* Adult participants >= 18 years with pathology confirmed any KSHV-positive aggressive B cell lymphomas, such as primary effusion lymphoma, and KSHV-associated large cell lymphoma
* Lymphoma that is measurable or assessable
* Any HIV status
* Hematologic and biochemical parameters within pre-specified limits at screening
* Willing to use effective birth control, as defined in the full protocol
* Neither pregnant nor breast feeding
* Excluded if other serious co-morbid condition that would prohibit administration of planned chemotherapeutic intervention is present

Design

* This is a phase I/ II study of lenalidomide in combination rituximab and modified DA-EPOCH (EPOCH-R^2) in participants with KSHV-positive aggressive B cell lymphomas.
* Phase I of the study will evaluate lenalidomide 25 mg days 1-10 in combination with modified DA-EPOCH-R to determine safety and tolerability. Dose de-escalation doses of lenalidomide are 20 mg and 15 mg.
* Participants with HIV will generally be prescribed cART.
* In phase I, with up to 3 dose levels, 6-18 participants will be accrued (3-6 participants per level).
* In the phase II portion of the study, 15 evaluable participants will be enrolled over 48-60 months and 12 months follow-up after the last participant has enrolled, a 1-tailed 0.10 alpha level test would have 80% power to determine if overall survival (OS) curve would demonstrate a 1-year OS consistent with 45% or better and ruling out 20% or worse.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Any Kaposi sarcoma herpesvirus (KSHV)-positive aggressive B cell lymphomas, such as primary effusion lymphoma (PEL), and KSHV-associated large cell lymphoma that is pathologically confirmed by the National Cancer Institute (NCI) Laboratory of Pathology
* Measurable or assessable lymphoma.
* Any human immunodeficiency virus (HIV) status
* Age 18 years or greater. Because no dosing or adverse event data are currently available on the use of lenalidomide in combination with etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin, and rituximab (EPOCH-R) in participants <18 years of age, children are excluded from this study but may be eligible for future pediatric trials.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-4.
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 14 days prior to and again within 1 day before starting lenalidomide and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide. Females of reproductive potential must adhere to the scheduled pregnancy testing as required in the Revlimid Risk Evaluation and Mitigation Strategy (REMS) program. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a vasectomy. All subjects must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure. Risks of Fetal Exposure, Pregnancy Testing Guidelines and Acceptable Birth Control
* All study participants must agree to be registered into the mandatory REVLIMID REMS program, and be willing and able to comply with the requirements of the REVLIMID REMS program.
* Able to take aspirin 81mg orally daily or if intolerant of aspirin, able to take a substitute thromboprophylaxis such as low molecular weight heparin.
* Ability of subject to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* Use of other systemic anticancer treatments or agents within the past 2 weeks. The use of rituximab for the treatment of KSHV-associated multicentric Castleman disease (MCD) or KSHV inflammatory cytokine syndrome (KICS) or the use of steroids are allowed within 2 weeks prior to start of treatment.
* Phase I or Phase II participants who have received prior dose-adjusted EPOCH for treatment for PEL or KSHV-associated large cell lymphoma
* Phase II participants who have received any prior curative-intent therapy for PEL or KSHV-associated large cell lymphoma. Participants who have received prior treatment as a bridge to curative-intent therapy will be considered per PI discretion.
* Parenchymal brain involvement with lymphoma
* History of malignant tumors other than KS or KSHV-associated MCD, unless:

  * In complete remission for greater than or equal to 1 year from the time response was first documented or
  * Completely resected basal cell carcinoma or
  * In situ squamous cell carcinoma of the cervix or anus
* Inadequate renal function, defined as calculated or estimated creatinine clearance < 60 mL/min unless lymphoma, KSHV-MCD, or KICS- related for calculation of creatinine clearance)
* Inadequate hepatic function
* Bilirubin (total) > 1.5 times the upper limit of normal; aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) > 3 times the upper limit of normal; EXCEPTIONS:

  * Total bilirubin greater than or equal to 5 mg/dL in participants with Gilbert's syndrome as defined by >80% unconjugated
  * Total bilirubin greater than or equal to 7.5 with direct fraction > 0.7 if participants is receiving a protease inhibitor at the time of initial evaluation
  * Hepatic dysfunction attributed to lymphoma, KSHV-MCD, or KICS
* Absolute neutrophil count (ANC) <1000/mm^3 and platelets < 75,000/mm^3 unless lymphoma, KSHV-MCD, or KICS- related.
* Common Terminology Criteria for Adverse Events (CTCAE)v5.0 Grade 3-4 neuropathy
* Ejection fraction less than 40% by echocardiography
* Known drug-related, inherited, or acquired procoagulant disorder including prothrombin gene mutation 20210, antithrombin III deficiency, protein C deficiency, protein S deficiency and antiphospholipid syndrome but not including heterozygosity for the Factor V Leiden mutation or the presence of a lupus anticoagulant in the absence of other criteria for the antiphospholipid syndrome.
* History of hypersensitivity reactions attributed to thalidomide, lenalidomide, or pomalidomide, including prior development of erythema nodosum if characterized by a desquamating rash while taking thalidomide, lenalidomide, or pomalidomide.
* Breast feeding (if lactating, must agree not to breast feed while taking lenalidomide). Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with lenalidomide, breastfeeding should be discontinued if the mother is treated with lenalidomide.
* Uncontrolled severe intercurrent illness including, but not limited to bacterial, fungal, or life-threatening viral infection; symptomatic congestive heart failure; unstable angina pectoris; cardiac arrhythmia; or psychiatric illness/social situations that would limit compliance with study requirements. Participants with severe intercurrent illnesses attributed to lymphoma, KSHV-MCD, or KICS may be eligible per principal investigators (PI's) or designees' discretion.
* Any condition, including laboratory abnormalities, which in the opinion of the Principal Investigator or Lead Associate Investigator, would prohibit administration of planned chemotherapeutic intervention, places the subject at unacceptable risk if they were to participate in the study or confounds the ability to interpret data from the study
* Pregnant women are excluded from this study because lenalidomide is a Category X agent with the potential for teratogenic or abortifacient effects. These potential risks may also apply to other agents used in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-07-03 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2027-10-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ramya Ramaswami, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI).

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2016-C-0171.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Lenalidomide+Etoposide Phosphate, Prednisone, Vincristine, Cyclophosphamide, Doxorubicin & Rituximab: Cohort 1, Dose Level 1 - Lenalidomide 25mg by mouth (PO) was given on days 1 to 10, plus, etoposide phosphate, prednisone, vincristine, cyclophosphamide, doxorubicin, and rituximab (DA-EPOCH-R). During cycle 1, Etoposide 50mg/m^2/day, Vincristine 0.4 mg/m^2 /day, and Doxorubicin 10 mg /m^2/day were given as continuous intravenous infusion days 6 to 9. During cycles 2-6, Etoposide, Vincristine 0.4 mg/m^2 /day, and Doxorubicin were given as continuous intravenous infusion days 1 to 4. During cycles 2-6, doses of etoposide and doxorubicin were adjusted based on hematologic parameters during the previous cycle. During cycle 1, Prednisone 60 mg/m^2 /day PO days 6 to 10. During cycles 2-6, Prednisone 60 mg/m^2 /day PO days 1-5. During cycle 1, Cyclophosphamide 750 mg/m^2 was given on day 10. During cycles 2-6, Cyclophosphamide 750 mg/m^2 was given on day 5. Rituximab was administered on day 4 prior to the start of EPOCH during cycle 1 and on day 1 during cycles 2 to 6.
Period: Phase I - Safety & Tolerability
Arm/Group | Lenalidomide+Etoposide Phosphate, Prednisone, Vincristine, Cyclophosphamide, Doxorubicin & Rituximab
Started | 6
Received Specified Dose | 6
Underwent Screening/Staging | 6
Evaluated for Response | 6
Off Treatment | 6
Off Study | 6
Disease Progression on Study | 1
Completed | 5
Not Completed | 1
Not completed — Did not complete last cycle of EPOCH-R2 due to progressive disease. | 1
Period: Phase II - Recommended Phase 2 Dose
Arm/Group | Lenalidomide+Etoposide Phosphate, Prednisone, Vincristine, Cyclophosphamide, Doxorubicin & Rituximab
Started | 11
Received Specified Dose | 11
Evaluated for Response | 11
Off Treatment | 11
Off Study | 11
Disease Progression on Study | 3
Completed | 7
Not Completed | 4
Not completed — Refused further treatment | 1
Not completed — Physician Decision | 2
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Lenalidomide+Etoposide Phosphate, Prednisone, Vincristine, Cyclophosphamide, Doxorubicin & Rituximab
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.53 (13.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 13
  White | 3
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: (Phase I) Maximum Tolerated Dose (MTD) of Etoposide, Prednisone, Vincristine, Cyclophosphamide, Doxorubicin, and Rituximab (DA-EPOCH-R2)
Description: The MTD is the dose level at which no more than 1 of up to 6 participants experiences dose-limiting toxicity (DLT) during the first two cycles of DA-EPOCH-R2 treatment. Association of treatment regimen with one-year overall survival.
  DLT is defined as any grade 4 adverse event at least possibly related to lenalidomide and not probably or definitely related to human immunodeficiency virus (HIV) or a Kaposi sarcoma-associated herpesvirus KSHV-associated malignancy resulting in a dose delay in etoposide phosphate, prednisone, vincristine, cyclophosphamide, doxorubicin, and rituximab (DA-EPOCH-R) treatment >2 weeks due to failure to resolve to grade 3 or lower. Any grade 3 cardiac toxicity that is at least possibly related to lenalidomide and not probably or definitely related to HIV or a Kaposi sarcoma-associated herpesvirus (KSHV)-associated malignancy resulting in a dose delay in DA-EPOCH-R treatment >2 weeks due to failure to resolve to grade 2 or lower.
Time Frame: First 6 weeks of treatment (2 cycles of treatment)
Population: 6/17 participants were analyzed because MTD was only assessed during phase I which was only 6 participants.
Measure: Number; unit: mg/day
Groups:
- All Participants: Cohort 1, Dose Level 1 - Lenalidomide 25mg by mouth (PO) was given on days 1 to 10, plus, etoposide phosphate, prednisone, vincristine, cyclophosphamide, doxorubicin, and rituximab (DA-EPOCH-R). During cycle 1, Etoposide 50mg/m^2/day, Vincristine 0.4 mg/m^2 /day, and Doxorubicin 10 mg /m^2/day were given as continuous intravenous infusion days 6 to 9. During cycles 2-6, Etoposide, Vincristine 0.4 mg/m^2 /day, and Doxorubicin were given as continuous intravenous infusion days 1 to 4. During cycles 2-6, doses of etoposide and doxorubicin were adjusted based on hematologic parameters during the previous cycle. During cycle 1, Prednisone 60 mg/m^2 /day PO days 6 to 10. During cycles 2-6, Prednisone 60 mg/m^2 /day PO days 1-5. During cycle 1, Cyclophosphamide 750 mg/m^2 was given on day 10. During cycles 2-6, Cyclophosphamide 750 mg/m^2 was given on day 5. Rituximab was administered on day 4 prior to the start of EPOCH during cycle 1 and on day 1 during cycles 2 to 6.
Arm/Group | All Participants
Number analyzed (Participants) | 6
mg/day | 25

2. Primary Outcome: (Phase II) Overall Survival in Treatment-naive Participants With Primary Effusion Lymphoma Treated With Etoposide, Prednisone, Vincristine, Cyclophosphamide, Doxorubicin, and Rituximab (DA-EPOCH-R2) Reported Along With a 90% Confidence Interval
Description: Median amount of time subject survives post therapy
Time Frame: End of follow up period (5 years)
Measure: Median (90% Confidence Interval); unit: years
Arm/Group | Lenalidomide+Etoposide Phosphate, Prednisone, Vincristine, Cyclophosphamide, Doxorubicin & Rituximab
Number analyzed (Participants) | 17
years | NA [0.40 to NA] — Median survival was not calculable because at the end of the follow-up period, more than 50% of the participants were still alive.

3. Primary Outcome: (Phase II) Overall Survival in Treatment-naive Participants With Primary Effusion Lymphoma Treated With Etoposide, Prednisone, Vincristine, Cyclophosphamide, Doxorubicin, and Rituximab (DA-EPOCH-R2) Reported Along With a 95% Confidence Interval
Description: Median amount of time subject survives post therapy.
Time Frame: End of follow up period (5 years)
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Lenalidomide+Etoposide Phosphate, Prednisone, Vincristine, Cyclophosphamide, Doxorubicin & Rituximab
Number analyzed (Participants) | 17
years | NA [0.36 to NA] — Median survival was not calculable because at the end of the follow-up period, more than 50% of the participants were still alive.

4. Secondary Outcome: Response Rate for Primary Effusion Lymphoma Reported Using a 90% Confidence Interval
Description: Response rate is defined as the percentage of participants who have either a complete response (CR) or partial response (PR) for primary effusion lymphoma treated with etoposide phosphate, prednisone, vincristine, cyclophosphamide, doxorubicin, and rituximab (DA-EPOCH-R2) measured by the International Working Group Response Criteria for Malignant Lymphomas. Complete response (CR) is complete disappearance of all detectable evidence of disease. Partial response (PR) is at least a ≥50% decrease in the sum of the product of the diameters of up to 6 of the largest dominant nodes or nodal masses.
Time Frame: Response rate was calculated at the end of treatment (18 weeks of treatment)
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Lenalidomide+Etoposide Phosphate, Prednisone, Vincristine, Cyclophosphamide, Doxorubicin & Rituximab
Number analyzed (Participants) | 17
percentage of participants | 76 [54 to 92]

5. Secondary Outcome: Response Rate for Primary Effusion Lymphoma Reported Using a 95% Confidence Interval
Description: as for outcome 4
Time Frame: Response rate was calculated at the end of treatment (after 18 weeks of treatment)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lenalidomide+Etoposide Phosphate, Prednisone, Vincristine, Cyclophosphamide, Doxorubicin & Rituximab
Number analyzed (Participants) | 17
percentage of participants | 76 [50 to 93]

6. Secondary Outcome: Progression-free Survival (PFS) for Primary Effusion Lymphoma Treated With Etoposide, Prednisone, Vincristine, Cyclophosphamide, Doxorubicin, and Rituximab (DA-EPOCH-R2) Using a 90% Confidence Interval
Description: PFS is defined as the duration of time from start of treatment to time of progression of Kaposi sarcoma-associated herpesvirus (KSHV)-lymphoma or death, whichever occurs first, measured by the International Working Group Response Criteria for Malignant Lymphoma. Progressive disease is appearance of any new nodal lesion ≥1.6 cm in greatest transverse diameter (GTD) or ≥1.1 cm in short axis during or after the end of therapy, even if other lesions are decreasing in size. At least a 50% increase from the nadir in the sum of the product of the diameters (SPD) of any previously involved nodes, or in a single involved node, or in the size of other lesions (e.g., splenic or hepatic nodules).
Time Frame: Over follow-up period, a median of 26 months
Measure: Median (90% Confidence Interval); unit: years
Arm/Group | Lenalidomide+Etoposide Phosphate, Prednisone, Vincristine, Cyclophosphamide, Doxorubicin & Rituximab
Number analyzed (Participants) | 17
years | 0.72 [0.37 to NA] — Upper end of the confidence interval of the Kaplan-Meier survival curve was not calculable because the proportion of participants who had progressive disease was too small.

7. Secondary Outcome: Progression-free Survival (PFS) for Primary Effusion Lymphoma Treated With Etoposide, Prednisone, Vincristine, Cyclophosphamide, Doxorubicin, and Rituximab (DA-EPOCH-R2) Using a 95% Confidence Interval
Description: as for outcome 6
Time Frame: Over a follow-up period, a median of 26 months
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | All Participants
Number analyzed (Participants) | 17
years | 0.72 [0.31 to NA] — Upper end of the confidence interval of the Kaplan-Meier survival curve was not calculable because the proportion of participants who had progressive disease was too small.

8. Secondary Outcome: Event-free Survival (EFS) for Primary Effusion Lymphoma Treated With Etoposide, Prednisone, Vincristine, Cyclophosphamide, Doxorubicin, and Rituximab (DA-EPOCH-R2) Reported Along With a 90% Confidence Interval
Description: Event-Free Survival (EFS) is defined as the duration of time from start of treatment to time of progression of Kaposi sarcoma-associated herpesvirus (KSHV)-lymphoma. Progressive disease was measured by the International Working Group Response Criteria for Malignant Lymphoma. Progressive disease is the appearance of any new nodal lesion ≥1.6 cm in greatest transverse diameter (GTD) or ≥1.1 cm in short axis during or after the end of therapy, even if other lesions are decreasing in size. At least a 50% increase from the nadir in the sum of the product of the diameters (SPD) of any previously involved nodes, or in a single involved node, or in the size of other lesions (e.g., splenic or hepatic nodules).
Time Frame: Over a follow-up period, a median of 26 months
Measure: Median (90% Confidence Interval); unit: years
Arm/Group | Lenalidomide+Etoposide Phosphate, Prednisone, Vincristine, Cyclophosphamide, Doxorubicin & Rituximab
Number analyzed (Participants) | 17
years | 0.72 [0.37 to NA] — Upper end of the confidence interval of the Kaplan-Meier survival curve was not calculable because the proportion of participants who had progressive disease was too small.

9. Secondary Outcome: Event-free Survival (EFS) for Primary Effusion Lymphoma Treated With Etoposide, Prednisone, Vincristine, Cyclophosphamide, Doxorubicin, and Rituximab (DA-EPOCH-R2) Reported Along With a 95% Confidence Interval
Description: as for outcome 8
Time Frame: Over a follow-up period, a median of 26 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lenalidomide+Etoposide Phosphate, Prednisone, Vincristine, Cyclophosphamide, Doxorubicin & Rituximab
Number analyzed (Participants) | 17
Months | 0.72 [0.31 to NA] — Upper end of the confidence interval of the Kaplan-Meier survival curve was not calculable because the proportion of participants who had progressive disease was too small.

10. Secondary Outcome: Response Assessment of Kaposi Sarcoma Using the Modified Acquired Immunodeficiency Syndrome (AIDS) Clinical Trials Criteria Reported Along With a 90% Confidence Interval
Description: Response was assessed by the percentage of participants with either a partial or complete response. Response was assessed using the Modified Acquired Immunodeficiency Syndrome (AIDS) Clinical Trials Criteria. Complete Response is the absence of any detectable residual disease, including tumor associated edema, persisting for at least 4 weeks. The absence of any detectable residual disease, including tumor associated edema, persisting for at least 4 weeks. Partial Response is a 50% or greater decrease in the number and/or size of previously existing lesions lasting for at least 4 weeks or no new lesions occurring in previously uninvolved areas of the body.
Time Frame: At end of treatment (after 18 weeks treatment)
Population: 4/17 participants were analyzed because only 4 participants had evaluable Kaposi sarcoma.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Lenalidomide+Etoposide Phosphate, Prednisone, Vincristine, Cyclophosphamide, Doxorubicin & Rituximab
Number analyzed (Participants) | 4
percentage of participants | 25 [1 to 75]

11. Secondary Outcome: Response Assessment of Kaposi Sarcoma Using the Modified Acquired Immunodeficiency Syndrome (AIDS) Clinical Trials Criteria Reported Along With a 95% Confidence Interval
Description: as for outcome 10
Time Frame: At end of treatment (after 18 weeks of treatment)
Population: 4/17 participants were analyzed because only 4 participants had evaluable Kaposi sarcoma.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lenalidomide+Etoposide Phosphate, Prednisone, Vincristine, Cyclophosphamide, Doxorubicin & Rituximab
Number analyzed (Participants) | 4
percentage of participants | 25 [0 to 81]

12. Secondary Outcome: Response Rate of Participants With Active Multicentric Castleman Disease (MCD) Assessed by the National Cancer Institute (NCI) MCD Response Criteria Reported Along With a 90% Confidence Interval
Description: Response rate is calculated by the percentage of participants with either a partial or complete response. Complete Response (CR) is full resolution of all clinical symptoms and laboratory abnormalities (whether or not these are indicator abnormalities) probably or definitely attributable to MCD, lasting at least 3 weeks. Partial Response (PR) is at least 50% of the abnormalities probably or definitely attributed to Kaposi sarcoma-associated herpesvirus (KSHV)-MCD must improve by the minimum amounts specified to attain PR (e.g., C-reactive protein reduction to ≤50% of baseline; and Hemoglobin increment 2g/dL not explained by transfusion).
Time Frame: At end of treatment (after 18 weeks of treatment)
Population: 5/17 participants were analyzed because responses were only measured in participants with MCD.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Lenalidomide+Etoposide Phosphate, Prednisone, Vincristine, Cyclophosphamide, Doxorubicin & Rituximab
Number analyzed (Participants) | 5
percentage of participants | 60 [19 to 92]

13. Secondary Outcome: Response Rate of Participants With Active Multicentric Castleman Disease (MCD) Assessed by the National Cancer Institute (NCI) MCD Response Criteria Reported Along With a 95% Confidence Interval
Description: as for outcome 12
Time Frame: At end of treatment (after 18 weeks of treatment)
Population: 5/17 participants were analyzed because responses were only measured in participants with MCD.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lenalidomide+Etoposide Phosphate, Prednisone, Vincristine, Cyclophosphamide, Doxorubicin & Rituximab
Number analyzed (Participants) | 5
percentage of participants | 60 [15 to 95]

14. Secondary Outcome: Kaposi's Sarcoma-associated Herpesvirus (KSHV)-Associated Inflammatory Cytokine Syndrome (KICS) Reported Along With a 90% Confidence Interval
Description: Complete Response (CR) is full resolution of all clinical symptoms and laboratory abnormalities (whether or not these are indicator abnormalities) probably or definitely attributable to KICS, lasting at least 3 weeks. Partial Response (PR) is at least 50% of the abnormalities probably or definitely attributed to KICS must improve by the minimum amounts (e.g., C-reactive protein reduction to ≤50% of baseline; and Hemoglobin increment 2g/dL not explained by transfusion). Progressive disease (PD) is at least two indicator abnormalities must deteriorate by the minimum amounts specified below to constitute PD (e.g., C-reactive protein increase by ≥50% of baseline (or the upper limit of normal, whichever is greater); Hemoglobin decrement 2g/dL not otherwise explained; and Platelet decrement ≥25,000/mm^3 not otherwise explained). Stable disease (SD) is no change in signs and symptoms of KICS that meet criteria for any of CR, PR or PD.
Time Frame: At the end of treatment (after 18 weeks of treatment)
Population: This outcome was not done because the definition of KSHV-inflammatory Cytokine syndrome (KICS) has been updated to exclude participants with lymphoma and therefore, effect of the regimen on KICS cannot be performed.
Arm/Group | Lenalidomide+Etoposide Phosphate, Prednisone, Vincristine, Cyclophosphamide, Doxorubicin & Rituximab
Number analyzed (Participants) | 0

15. Secondary Outcome: Kaposi's Sarcoma-associated Herpesvirus (KSHV)-Associated Inflammatory Cytokine Syndrome (KICS) Reported Along With a 95% Confidence Interval
Description: as for outcome 14
Time Frame: At the end of treatment (after 18 weeks of treatment)
Population: as for outcome 14
Arm/Group | Lenalidomide+Etoposide Phosphate, Prednisone, Vincristine, Cyclophosphamide, Doxorubicin & Rituximab
Number analyzed (Participants) | 0

16. Secondary Outcome: Pharmacokinetics of Lenalidomide in Blood
Description: Bioanalytical measurements will be conducted on an ultra-high-performance liquid chromatography (uHPLC) with tandem mass spectrometric detection to determine the concentration of lenalidomide in blood using an assay developed and validated by the National Institutes of Health (NIH) Clinical Pharmacology Program.
Time Frame: Cycle 1 Day 1(C1D1), C1D7, C6D1 (one cycle = 21 days)
Reporting Status: Not Posted, anticipated posting 2026-12

17. Secondary Outcome: Pharmacokinetics of Lenalidomide Effusion
Description: Bioanalytical measurements will be conducted on an ultra-high-performance liquid chromatography (uHPLC) with tandem mass spectrometric detection to determine the concentration of lenalidomide in effusions using an assay developed and validated by the National Institutes of Health (NIH) Clinical Pharmacology Program.
Time Frame: Cycle 1 Day 1(C1D1), C1D7, C6D1 (one cycle = 21 days)
Population: The objective of obtaining effusion-based PKs can only be done if effusions within a cavity are visible after treatment and safe to proceed. Safety is paramount in this Phase I study and therefore if there was no effusion and/or if it was not safe to sample based on investigator judgement, no samples could be obtained, and no PKs could be obtained to answer this objective. There is no data collected for this measure of effusion PKs.
Arm/Group | Lenalidomide+Etoposide Phosphate, Prednisone, Vincristine, Cyclophosphamide, Doxorubicin & Rituximab
Number analyzed (Participants) | 0

18. Secondary Outcome: Pharmacokinetics of Lenalidomide in Cerebrospinal Fluid (CSF)
Description: Bioanalytical measurements will be conducted on an ultra-high-performance liquid chromatography (uHPLC) with tandem mass spectrometric detection to determine the concentration of lenalidomide in CSF using an assay developed and validated by the National Institutes of Health (NIH) Clinical Pharmacology Program.
Time Frame: Cycle 1 Day 1(C1D1), C1D7, C6D1 (one cycle = 21 days)
Reporting Status: Not Posted, anticipated posting 2026-12

19. Other Pre Specified Outcome: Number of Participants With a Dose-limiting Toxicity (DLT)
Description: DLT's as assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). DLT is defined as any grade 4 adverse event at least possibly related to lenalidomide and not probably or definitely related to human immunodeficiency virus (HIV) or a Kaposi sarcoma-associated herpesvirus (KSHV)associated malignancy resulting in a dose delay in etoposide phosphate, prednisone, vincristine, cyclophosphamide, doxorubicin, and rituximab (DA-EPOCH-R) treatment >2 weeks due to failure to resolve to grade 3 or lower. Any grade 3 cardiac toxicity that is at least possibly related to lenalidomide and not probably or definitely related to HIV or a KSHV-associated malignancy resulting in a dose delay in DA-EPOCH-R treatment >2 weeks due to failure to resolve to grade 2 or lower. DLT's were used to determine whether to stop or hold therapy in an individual participant as well as to expand individual dose levels from 3 to 6 participants.
Time Frame: First 6 weeks (2 cycles) of treatment
Population: 6/17 participants were analyzed because dose-limiting toxicity was only performed during phase I which was only 6 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Lenalidomide+Etoposide Phosphate, Prednisone, Vincristine, Cyclophosphamide, Doxorubicin & Rituximab
Number analyzed (Participants) | 6
Participants | 0

20. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Median follow-up time was 26 months
Measure: Count of Participants; unit: Participants
Arm/Group | Lenalidomide+Etoposide Phosphate, Prednisone, Vincristine, Cyclophosphamide, Doxorubicin & Rituximab
Number analyzed (Participants) | 17
Participants | 17

ADVERSE EVENTS:
Time Frame: All-Cause Mortality was monitored/assessed for a median or 26 months. Adverse Events was monitored/assessed from the first study treatment through 30 days after the study agent (s) was/were administered.
Arm/Group | Lenalidomide+Etoposide Phosphate, Prednisone, Vincristine, Cyclophosphamide, Doxorubicin & Rituximab
All-Cause Mortality (participants affected / at risk) | 3/17
Serious Adverse Events (participants affected / at risk) | 12/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenalidomide+Etoposide Phosphate, Prednisone, Vincristine, Cyclophosphamide, Doxorubicin & Rituximab (N=17)
Abdominal pain (Gastrointestinal disorders) | 1 (2)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Chills (General disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Disease progression (General disorders) | 3 (3)
Dizziness (Nervous system disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Enterocolitis (Infections and infestations) | 1 (1)
Fatigue (General disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 8 (14)
Fever (General disorders) | 2 (6)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Hypotension (Vascular disorders) | 3 (3)
Hypothermia (General disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (2)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sepsis (Infections and infestations) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 2 (2)
Typhlitis (Gastrointestinal disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 1 (1)
Vascular disorders - Other, DVT upper extremities, bilateral (Vascular disorders) | 1 (1)
Vascular disorders - Other, Pulmonary emboly, LUL (Vascular disorders) | 1 (1)
Vascular disorders - Other, Pulmonary emboly, RLL (Vascular disorders) | 1 (1)
White blood cell decreased (Investigations) | 1 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenalidomide+Etoposide Phosphate, Prednisone, Vincristine, Cyclophosphamide, Doxorubicin & Rituximab (N=17)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Activated partial thromboplastin time prolonged (Investigations) | 1 (3)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (3)
Alanine aminotransferase increased (Investigations) | 7 (23)
Alkaline phosphatase increased (Investigations) | 7 (26)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (6)
Anal pain (Gastrointestinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 16 (242)
Anorexia (Metabolism and nutrition disorders) | 7 (10)
Anxiety (Psychiatric disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4)
Aspartate aminotransferase increased (Investigations) | 9 (28)
Atrial flutter (Cardiac disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4)
Blood bilirubin increased (Investigations) | 6 (18)
Blood lactate dehydrogenase increased (Investigations) | 2 (3)
Blurred vision (Eye disorders) | 1 (1)
CD4 lymphocytes decreased (Investigations) | 15 (43)
CPK increased (Investigations) | 7 (11)
Cardiac arrest (Cardiac disorders) | 1 (1)
Cardiac disorders - Other, specify: Tachycardia (Cardiac disorders) | 1 (1)
Cardiac disorders - Other, specify: shock (Cardiac disorders) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Cholesterol high (Investigations) | 6 (8)
Colitis (Gastrointestinal disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1)
Constipation (Gastrointestinal disorders) | 9 (12)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Creatinine increased (Investigations) | 8 (20)
Depression (Psychiatric disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 5 (7)
Dizziness (Nervous system disorders) | 1 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (6)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 3 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Dysuria (Renal and urinary disorders) | 1 (2)
Ear and labyrinth disorders - Other, specify: Ear infection (Ear and labyrinth disorders) | 1 (1)
Edema limbs (General disorders) | 4 (6)
Edema trunk (General disorders) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (4)
Esophagitis (Gastrointestinal disorders) | 2 (2)
Eye disorders - Other, specify: Photophobia (Eye disorders) | 1 (1)
Fatigue (General disorders) | 13 (33)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3)
Fever (General disorders) | 8 (17)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, specify: Gastric obstruction (Gastrointestinal disorders) | 1 (1)
General disorders and administration site conditions - Other, specify: Body aches (General disorders) | 1 (1)
General disorders and administration site conditions - Other, specify: Burning top of the feet (General disorders) | 1 (1)
General disorders and administration site conditions - Other, specify: Facial rash (General disorders) | 1 (1)
General disorders and administration site conditions - Other, specify: Imbalance (General disorders) | 1 (1)
General disorders and administration site conditions - Other, specify: Left Knee effusion (General disorders) | 1 (1)
General disorders and administration site conditions - Other, specify: Nodule, right breast (General disorders) | 1 (1)
General disorders and administration site conditions - Other, specify: Rash forehead (General disorders) | 1 (1)
General disorders and administration site conditions - Other, specify: Runny nose (General disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Headache (Nervous system disorders) | 6 (14)
Hematuria (Renal and urinary disorders) | 1 (1)
Hot flashes (Vascular disorders) | 1 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 8 (9)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (2)
Hypernatremia (Metabolism and nutrition disorders) | 4 (5)
Hyperphosphatemia (Metabolism and nutrition disorders) | 5 (8)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 14 (25)
Hyperuricemia (Metabolism and nutrition disorders) | 6 (10)
Hypoalbuminemia (Metabolism and nutrition disorders) | 15 (43)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 16 (71)
Hypomagnesemia (Metabolism and nutrition disorders) | 6 (12)
Hyponatremia (Metabolism and nutrition disorders) | 14 (40)
Hypophosphatemia (Metabolism and nutrition disorders) | 5 (8)
Hypotension (Vascular disorders) | 3 (4)
Hypothyroidism (Endocrine disorders) | 3 (5)
Infections and infestations - Other, specify: CMV viremia (Infections and infestations) | 1 (1)
Infections and infestations - Other, specify: Epiglottitis (Infections and infestations) | 1 (1)
Injury, poisoning and procedural complications - Other, specify: DVT-LUA axillary/basilica vein (Injury, poisoning and procedural complications) | 1 (1)
Insomnia (Psychiatric disorders) | 4 (7)
Lymphocyte count decreased (Investigations) | 17 (306)
Malaise (General disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 7 (16)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Nail discoloration (Skin and subcutaneous tissue disorders) | 5 (6)
Nausea (Gastrointestinal disorders) | 10 (21)
Neutrophil count decreased (Investigations) | 17 (191)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Oral pain (Gastrointestinal disorders) | 3 (3)
Pain (General disorders) | 8 (14)
Paresthesia (Nervous system disorders) | 1 (1)
Periorbital edema (Eye disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 2 (4)
Peripheral sensory neuropathy (Nervous system disorders) | 9 (29)
Platelet count decreased (Investigations) | 17 (174)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (8)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 9 (13)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (5)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3)
Renal and urinary disorders - Other, specify: Uric acid increased (Renal and urinary disorders) | 1 (1)
Renal and urinary disorders - Other, specify: Urine protein increased (Renal and urinary disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Respiratory, thoracic and mediastinal disorders - Other, specify: Runny nose (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sepsis (Infections and infestations) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 2 (3)
Sinusitis (Infections and infestations) | 2 (2)
Skin and subcutaneous tissue disorders - Other, specify: Brittle nails (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify: Darkening of skin (Skin and subcutaneous tissue disorders) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (2)
Skin infection (Infections and infestations) | 2 (3)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thrush (Infections and infestations) | 2 (2)
Upper respiratory infection (Infections and infestations) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (4)
Vascular disorders - Other, specify: Pulmonary emboly, LUL (Vascular disorders) | 1 (3)
Vascular disorders - Other, specify: Pulmonary emboly, RLL (Vascular disorders) | 1 (3)
Vomiting (Gastrointestinal disorders) | 4 (4)
Weight loss (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 17 (274)
Weight loss (Investigations) | 0 (0)
White blood cell decreased (Investigations) | 1 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-06-06): https://cdn.clinicaltrials.gov/large-docs/42/NCT02911142/Prot_SAP_000.pdf
  • Informed Consent Form (2023-08-01): https://cdn.clinicaltrials.gov/large-docs/42/NCT02911142/ICF_001.pdf